CLINICAL TRIAL: NCT05116475
Title: Evaluation of dAroLutamide Addition to anDrogen Deprivation Therapy and radIatioN Therapy in Newly Diagnosed Prostate Cancer With Pelvic Lymph Nodes Metastases
Acronym: ALADDIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALADDIN
Record Dates: First submitted 2021-10-27; First posted 2021-11-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Darolutamide; ARTIC; Bayer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Arm A: ADT + Intensity-Modulated Image-Guided Radiation Therapy + Darolutamide ADT will be associated with LHRH agonists or antagonists for 24 months4. Darolutamide regimen will be of 2 tablets of 300 mg orally twice daily for 24 months.
  Interventions: Drug: Darolutamide 300 mg
- Arm B (Placebo Comparator): Arm B: ADT + Intensity-Modulated Image-Guided Radiation Therapy + Placebo of Darolutamide
  ADT will be associated with LHRH agonists or antagonists for 24 months4. Darolutamide regimen will be of 2 tablets of 300 mg orally twice daily for 24 months.
  Interventions: Drug: Placebo of Darolutamide

INTERVENTIONS:
Drug: Darolutamide 300 mg — Darolutamide regimen will be of 2 tablets of 300 mg orally twice daily for 24 months.
  Arms: Arm A
Drug: Placebo of Darolutamide — Placebo of Darolutamide regimen will be of 2 tablets of 300 mg orally twice daily for 24 months.
  Arms: Arm B

SUMMARY:
Prospective, multicenter, comparative, randomized placebo-controlled Phase III trial - patients with hormone-naïve prostate cancer and pelvic lymph nodes metastases

DETAILED DESCRIPTION:
Standard of care for patients with prostate cancer (PC) with pelvic lymph nodes metastases is radiotherapy (RT) with long-term androgen deprivation therapy (ADT). . Darolutamide improves survival in men with castration-refractory non metastatic prostate cancer. We hypothesize that adding Darolutamide to ADT and RT could improve FFS for these high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

1. . Newly diagnosed, histologically confirmed prostate adenocarcinoma
2. ≥ 18 years old.
3. Initial staging with Pelvic MRI, body CT-scan/bone scan or Choline or PSMA PET-CT
4. Any T stage
5. N stage: N1 - Pelvis lymph nodes metastases (upper limit defined as the L4/L5 interspace).
6. Intention to treat with long-term androgen deprivation therapy (24 months).
7. Hormonal therapy with LH-RH agonist or antagonist is allowed up to 3months prior to randomization.
8. Able to receive protocol therapy and have life expectancy of at least 36 months, ECOG Performance Status (PS) 0-2.
9. . Blood counts at screening: hemoglobin ≥ 9.0 g/dl, absolute neutrophil count ≥ 1500/μl (1.5x109/l), platelet count ≥ 100,000/μl (100x109/l ) (patient must not have received any growth factor or blood transfusion within 7 days of the hematology laboratory obtained at screening).
10. Screening values of serum alanine aminotransferase (ALT) and/or aspartate transaminase (AST) < 2.5 x upper limit of normal (ULN), total bilirubin < 1.5 x ULN (except patients with a diagnosis of Gilbert's disease), creatinine < 2.0 x ULN.
11. Sexually active patients, unless surgically sterile, must agree to use condoms as an effective barrier method during the study treatment and for 3 months after the end of the study treatment.
12. Written informed consent.
13. Willing and expected to comply with follow-up schedule.
14. Affiliated to the social security system.
15. Use of 5-α reductase inhibitors (finasteride, dutasteride) is allowed

Exclusion Criteria:

1. Lymph nodes metastases outside of the pelvis
2. Bone or visceral metastases
3. Prior systemic therapy for locally-advanced prostate cancer except for LH-RH agonist or antagonist up to 3 months before randomization
4. Prior treatment with:

   * Second generation AR inhibitors such as enzalutamide, apalutamide (ARN-509), darolutamide (ODM-201) other investigational AR inhibitors
   * CYP17 enzyme inhibitor such as abiraterone acetate, TAK-700 or
   * Oral ketoconazole
   * Use of estrogens, or AR inhibitors (bicalutamide, flutamide, nilutamide, cyproterone acetate)
5. Use of systemic corticosteroid with dose greater than the equivalent 10 mg of prednisone/day within 28 days before randomization.
6. Patients with QTor QTc interval > 450 ms on the ECG
7. Initiation of treatment with bisphosphonate or denosumab within 12 weeks before randomization. Patients receiving bone loss prevention treatment on a stable dose of e.g. bisphosphonate or denosumab for at least 28 days before randomization can continue the treatment during the study.
8. Known hypersensitivity to the study treatment (RT, ADT, darolutamide/placebo) or any of its ingredients.
9. Major surgery within 28 days before randomization.
10. Any of the following within 6 months before randomization: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft; congestive heart failure New York Heart Association (NYHA) Class III or IV or arterial thromboembolic event.
11. Uncontrolled hypertension as indicated by a resting systolic BP > 160 mmHg or diastolic BP > 100 mmHg at screening. Patients may be re-screened after adjustments of anti- hypertensive medications.
12. Prior malignancy. Adequately treated basal cell or squamous cell carcinoma of skin or superficial bladder cancer that has not spread behind the connective tissue layer (i.e. pTis, pTa, and pT1) is allowed, as well as any other cancer for which chemotherapy has been completed > 5 years ago and from which the patient has been disease-free.
13. Gastrointestinal disorder or procedure which expects to interfere significantly with absorption of study treatment.
14. Active viral hepatitis, active human immunodeficiency virus (HIV) or chronic liver disease.
15. Participation in another interventional clinical trial and any concurrent treatment with any investigational drug
16. Any condition that in the opinion of the investigator would impair the patients' ability to comply with the study procedures.
17. Unable to swallow study medications and comply with study requirements.
18. Galactose intolerance, the Lapp lactase deficiency or glucose galactose-malabsorption
19. History of bilateral hip replacements making IMRT impossible
20. Contra-indications for the administration of any of the study treatments (RT, ADT, Darolutamide/placebo) or any of its ingredients.
21. Patient under guardianship, administrative tutorship and incapable to give informed consent

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival FFS | 3 years
  The failure-free survival is defined as the time from the date of randomization to clinical (new cancer-related symptoms), biochemical (PSA rising) or radiological (local relapse or new metastases) progression, death, end of 3-year follow-up period or lost to follow-up, whichever occurs first.

SECONDARY OUTCOMES:
Metastasis-free survival rates | 3 years
  To evaluate the metastasis-free survival rates
Progression free survival rate | 3 years
  To evaluate the progression free survival rates
PSA response levels | 3 years
  PSA response is defined by the rate of patients having a decrease of > 50% of their PSA level, as measured every 3 months from the date of randomization to the date of a documented biochemical relapse.
Overall survival rates | 3 years
  Overall survival is defined as the time from the date of randomization to the date of documented death from any cause, end of 3-year follow-up period or lost to follow-up, whichever occurs first
Cancer-specific survival rates | 3 years
  Cancer-specific survival is defined as the time from the date of randomization to the date of documented death from prostate cancer or complication from the treatment, end of 3-year follow-up period or lost to follow-up, whichever occurs first
Time to pain progression | 3 years
  Time to pain progression is defined as the time from the date of randomization to the date of documented pain, end of 3-year follow-up period or lost to follow-up, whichever occurs first
Toxicities | 3 years
  To evaluate toxicities (CTCAE v5.0) due to treatements
Quality of life of the patient | 3 years
  Quality of life will be assessed using self-administered questionnaires (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire : EORTC QLQ-C30 v2)
Quality of life of the patient | 3 years
  Quality of life will be assessed using self-administered questionnaires (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire : EORC QLQ-PR25 V3)
Quality of life of the participants | 3 years
  Quality of life will be assessed using self-administered questionnaires (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire : EORTC QLQ-PR253) by patients

CONTACTS AND LOCATIONS:
Overall Officials: Pierre COMBE, MD, Principal Investigator — Centre Oncologie Radiothérapie 37 - CORT37
Locations (1):
- Pôle Santé Léonard de Vinci, Chambray-lès-Tours, France

IPD SHARING:
Plan to Share IPD: No